CLINICAL TRIAL: NCT04744857
Title: A Prospective，Multicenter, Single-arm Clinical Trial to Evaluate Safety and Efficacy of TaurusOne® Transcatheter Aortic Valve Replacement System With Retrievable Delivery Catheter System
Brief Title: Safety and Efficacy of TaurusOne® Transcatheter Aortic Valve Replacement System With Retrievable Delivery Catheter System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peijia Medical Technology (Suzhou) Co., Ltd. (Industry)
Collaborators: General Hospital of Shenyang Military Region (Other); Shanghai Zhongshan Hospital (Other); Guangdong Provincial People's Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Air Force Military Medical University, China (Other); West China Hospital (Other); Beijing Anzhen Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Central South University (Other); Fu Wai Hospital, Beijing, China (Other); China National Center for Cardiovascular Diseases (Other Government); Shanghai Lingsi Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP12001
Record Dates: First submitted 2021-01-29; First posted 2021-02-09 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Membrane Transport Proteins

STUDY DESIGN:
Intervention Model Description: Preliminary data from the TaurusOne® clinical trial show good safety and efficacy in this trial without altering the artificial aorta To evaluate the safety and effectiveness of a transporter with a recoverable function. Take TaurusOne® in a clinical trial of compounding Endpoint event incidence was used as a target control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single set of test (Experimental): The experimental apparatus consisted of artificial aortic valve, transporter and grip-loading system.
  Interventions: Combination Product: The experimental apparatus consisted of artificial aortic valve, transporter and grip-loading system.

INTERVENTIONS:
Combination Product: The experimental apparatus consisted of artificial aortic valve, transporter and grip-loading system. — Using the grip-loading system, the artificial aortic valve was squeezed and loaded into the sheath of the transporter through the vascular approach.The artificial aortic valve is delivered and positioned at the correct anatomical position for release. For example, the artificial main valve is displayed after partial release If the aortic valve is not in the correct anatomical position, the artificial aortic valve can be recovered and placed into the sheath tube of the transporter for re-positioning and release.
  Other Names: The TaurusOne® transcatheter aortic valve replacement system features a retrievable delivery catheter system

SUMMARY:
The TaurusOne® transcatheter aortic valve system with retrievable delivery catheter system is evaluated the safety and effectiveness for the delivery of artificial aortic valve in a prospective, multicenter, single-arm clinical trial.

DETAILED DESCRIPTION:
The TaurusOne® transcatheter aortic valve system with retrievable delivery catheter system is evaluated the safety and effectiveness for the delivery of artificial aortic valve in a prospective, multicenter, single-arm clinical trial. According to the inclusion and exclusion criteria, sixty patients are planed been enrolled and implanted with TaurusOne® .Patients are seen at pre and post procedure, discharge, 30 days. The main follow-up included clinical symptoms and signs, cardiac ultrasound, CT, etc. The outcome included immediate device success, procedure success, And the major cardiovascular and cerebrovascular adverse events (MACCE, including mortality, stroke, myocardial infarction, reoperation, arrhythmia, conduction block).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing to participate and sign the informed consent and can cooperate with the whole trial process;
* Age ≥70 years old;
* Patients with severe calcified aortic stenosis confirmed by echocardiography (trans-aortic valve flow velocity ≥ 4.0m /s, or trans-active valvular pressure difference ≥40mmHg (1mmHg=0.133kPa), or aortic valve orientation area < 0.8cm2, or effective aortic valve orifice the product index is < 0.5cm2/m2);
* Appear obvious symptoms caused by aortic stenosis, NYHA class Ⅱ or higher;
* The cardiac team (at least two specialists in cardiovascular surgery) assessed the patient as unsuitable for routine surgery ;
* The life expectancy of the patient after implantation of the prosthetic valve was evaluated by the cardiac team (at least two specialists in cardiovascular surgery) as more than one year;
* Patients with aortic ring diameter ≥18mm and ≤29mm (cardiac CT measurement);
* The diameter of the ascending aorta of the patient was < 50mm.

Exclusion Criteria:

* Patients with bacteremia or toxemia;
* previous history or active endocarditis;
* Acute myocardial infarction (Q-wave MI, or non-Q-wave MI with increased creatine kinase isoenzyme and/or troponin T) within 30 days;
* Echocardiography found any intracardiac mass, left ventricle or atrial thrombosis, vegetations;
* Symptomatic atrial fibrillation that cannot be improved by medication;
* Familial hypertrophic cardiomyopathy;
* Mitral valve and tricuspid valve insufficiency (reflux Ⅱ level above);
* Prior aortic valve grafts (mechanical or biological valve stents);
* Known allergy to contrast agent, aspirin, heparin, ticlopidine, nickel-titanium memory alloy, or bovine products;
* Known to be contraindication or allergic to all anticoagulant regimens, or unable to use anticoagulant during the test;
* Other serious diseases that may reduce life expectancy to less than 12 months (e.g. clinically recurrent or metastatic cancer, congestive heart failure, etc.)
* Current drug abuse problem (e.g., alcohol, cocaine, heroin, etc.); Plan to undergo surgery that may cause nonadherence to protocol or confusion in data interpretation.
* Cerebrovascular accident (CVA) in the past 6 months;
* Patients with common or internal carotid or vertebral artery stenosis (> 70%);
* WBC count < 3×109/L, platelet count < 50×109/ L;
* Hemoglobin < 90g/L;
* Patients with severe coagulation dysfunction;
* Severe left ventricular dysfunction, left ventricular ejection fraction < 20%;
* Abdominal or thoracic aortic aneurysm;
* Hepatic encephalopathy or acute active hepatitis;
* Receiving dialysis or a baseline creatinine level of > 3.0 mg/dL (266μmol/L);
* Have bleeding tendency or history of coagulation disease or refuse blood transfusion;
* Have active gastric ulcer or active gastrointestinal (GI) bleeding;
* Suffer from neurological diseases that seriously affect the ability to move or live in daily life;
* People with mental illness or mental disorder who cannot express themselves normally;
* Need emergency surgery for any reason;
* Screening participants who had participated in other drug or medical device clinical trials within the previous 3 months;
* Other conditions considered by the investigator to be inappropriate for participation in this clinical trial.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Composite event rate at 30 days | 30 days after procedure
  Patient-oriented composite event including all-cause death，severe stroke，myocardial infarction, permanent pacemaker implantation，surgical reoperation and valve-in-valve.

SECONDARY OUTCOMES:
Device success rate (immediately after procedure) | Immediately after procedure
  Device success is defined as
  * Vascular access, artificial aortic valve delivery and release were successful, and the delivery catheter was successfully withdrawn.
  * The artificial aortic valve was implanted in an anatomically accurate position.
  * The artificial aortic valve met the expected requirements (mean transvalvular pressure difference < 20mmHg or maximum flow rate < 3m/s; No serious manual initiative valve regurgitation or perivalvular leakage)
Procedure success rate | 72 hours after procedure/prior to discharge
  Procedure success is defined as the artificial aortic valve successfully implanted in the correct anatomical position 72h after surgery or before discharge without severe artificial aortic valve regurgitation or perivalvular leakage.
Cardiac function improvement | 30 days after procedure
  Cardiac function improvement is accessed by NYHA cardiac function classification increases from baseline to 30 days.
Quality of life of patients | 30 days after procedure
  Quality of Life of patients accessed by EuroQol-5 Dimensions (EQ-5D) Questionnaire. The higher scores mean a worse health state. Recording changes from baseline to 30 days.

OTHER OUTCOMES:
Product performance evaluation | Immediately after procedure
  Product Performance includes grip loading, emptying , delivery, release, retrace, development and retrieval performance of delivery catheter system. Every item measured by:1=good 2=average 3=poor.
operative complication | Immediately after procedure
  The rate of operative complication
The incidence of major adverse cardiovascular and cerebrovascular events during the trial(MACCEs) | 30 days after procedure
  Incidence of MACCEs (including mortality, stroke, myocardial infarction, and so on surgery, arrhythmias, conduction blocks) during the trial.
Incidence of major adverse valvular events (MAVREs) during the trial | 30 days after procedure
  Incidence of MAVREs (including artificial aortic valve-related death, permanent cardiac pacemaker or defibrillator implantation, artificial aortic valve embolism or thrombosis, artificial aortic valve loss of function) during the trial.
hemorrhage | 30 days after procedure
  Rate of patients with hemorrhage during the trial.
acute kidney injury | 30 days after procedure
  Rate of patients with acute kidney injury during the trial.
Other TAVI related complications | 30 days after procedure
  Rate of patients with Other TAVI related complications during the trial. Other TAVI related complications include conversion to surgery, accidental cardiopulmonary mechanical assistance, coronary occlusion, ventricular septal perforation, mitral valve damage or loss of function, pericardial tamponade, endocarditis, valvular thrombosis, valvular ectopic (displacement, embolization, erroneous release), etc.
Valvular function | 30 days after procedure
  Valvular function include valve stenosis, valve regurgitation, valve function (such as opening area, pressure gradient), perivalvular leakage, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Peiga Medical Technology (Suzhou) Co., Ltd, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No